CLINICAL TRIAL: NCT06469580
Title: Neonatologist-performed Lung Ultrasound (NPLUS) to Guide Respiratory Therapy to Prevent Extubation Failure in Term and Preterm Neonates- a Randomized Controlled Pilot Trial
Brief Title: Neonatologist-performed Lung Ultrasound (NPLUS) to Guide Respiratory Therapy to Prevent Extubation Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36-187 ex 23/24
Record Dates: First submitted 2024-05-21; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Neonatal Disease
Keywords: neonatologist performed lung ultrasound; extubation failure; neonates; consolidation
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPLUS group (Experimental): In the NPLUS group (intervention group) lung ultrasound is performed at time point T0 (prior to extubation), T1 (2-4 hours post extubation) and time point T2 (16-24 h) post extubation.
  Interventions: Other: NPLUS (neonatologist performed lung ultrasound)
- control group (No Intervention): Includes routine care in the control group in case of clinical (respiratory) deterioration which is optional chest x-ray or NPLUS at any time point after extubation indicated by the clinician in charge. There are no study-specific measures in the control group.

INTERVENTIONS:
Other: NPLUS (neonatologist performed lung ultrasound) — NPLUS is conducted with an ultrasound scanner using a high-frequency (12-15 MHz) linear transducer probe (scanning depth approximately 4-5 cm). The neonate is placed in a supine position. The anterior, lateral and posterior chest areas are scanned using the presets "lung" or "small parts". Landmarks are the anterior and posterior axillary line (longitudinal) on each hemithorax. A sequential scan from right to left, anterior to posterior is performed. (6 lung areas). In the study NPLUS is performed to quantify the lung ultrasound score at time points T0, T1 and T2. Sequences of 3-5 seconds are saved and assessed according to the lung ultrasound score adapted by Rodriguez-Fanjul et al. (0- to 3 point score for each area, resulting in a total score ranging from 0 to 18). To ensure inter-observer reliability the anonymous video sequences are then rated by two independent neonatologists.
  Arms: NPLUS group

SUMMARY:
The objective of the study is to evaluate the role of neonatologist-performed lung ultrasound (NPLUS) after weaning from invasive mechanical ventilation and extubation. Our aim is to study the diagnostic accuracy of NPLUS and investigate whether LUS leads to earlier actions before clinical deterioration and hence prevents extubation failure.

DETAILED DESCRIPTION:
In the past few years, lung ultrasound has been established as a tool to dynamically assess the lungs in various clinical conditions. Standardized protocols have been compiled to allow for an easy and fast evaluation. The point-of-care ultrasound (POCUS) is easily accessible and allows the clinician a readily available bed-side evaluation.

Although invasive mechanical ventilation displays a lifesaving strategy in neonatal intensive care, it is associated with numerous long-term complications especially in preterm infants. Despite a shift to lung-protective ventilation, time on mechanical ventilatory support should be kept as short as possible, considering timely weaning and switch to a non-invasive ventilation. Estimating the right time for discontinuation of invasive mechanical ventilation remains challenging and is influenced by several parameters. Extubation failure can be associated with respiratory failure following exhaustion on non-invasive ventilatory support.

Collapse of alveolar units lead to hypo-aerated areas. Small airway size, obstruction due to secretion and muscular weakness predispose to the development of atelectasis in neonates. Atelectasis occurring post extubation are a frequent cause of extubation failure. Lung consolidations can be sonographically detected. A sensitivity of 100% for the detection of neonatal pulmonary atelectasis has been described. In recent studies Lung Ultrasound Severity Score (LUSS) has been shown to be an independent predictor of successful extubation in mechanically ventilated preterm infants. However, once extubated, only limited data is available if extubation failure later in the process can be predicted. Lung aeration decreased after extubation to spontaneous breathing.

Early standardized evaluation of the lung via lung ultrasound can deliver important information on aeration of the lungs and whether action may be required. Using a standardized protocol (lung ultrasound score, LUS) on certain timepoints after extubation can lead to early detection of loss of aeration. Timely intervention with e.g., temporary PEEP increase for alveolar recruitment on non-invasive ventilatory support, positioning of the patient prior to clinical deterioration can impede the need of a reintubation and invasive mechanical ventilatory support.

ELIGIBILITY:
Inclusion Criteria:

* All preterm and full-term neonates receiving invasive mechanical ventilation at the Division of Neonatology of the Medical University of Graz AND
* Written informed consent was obtained from parents prior to extubation

Exclusion Criteria:

none

Ages: 1 Minute to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Reintubation rate (within 72 hours after extubation) | within 72 hours after extubation

SECONDARY OUTCOMES:
Mode of respiratory support | within 72 hours after extubation
  NCPAP, DUOPAP or BILEVEL during 72 hours after extubation
Respiratory settings- FiO2 | within 72 hours after extubation
  FiO2 (fraction of inspired oxygen) during 72 hours after extubation
Respiratory settings- PEEP | within 72 hours after extubation
  PEEP (Positive EndExpiratory Pressure) during 72 hours after extubation
SpO2/FiO2 ratio | every hour during 72 hours after extubation
  Ratio of arterial oxygen saturation and fraction of inspired oxygen
pH from capillary blood gas analysis | within 72 hours after extubation
  pH routinely obtained capillary blood gas analysis at certain time points within 72 hours after extubation
Carbon dioxide partial pressure (pCO2) | within 72 hours after extubation
  pCO2 Routinely obtained capillary blood gas analysis at certain time points within 72 hours after extubation
Base Excess (BE) | within 72 hours after extubation
  BE routinely obtained capillary blood gas analysis at certain time points within 72 hours after extubation
Number of lung imaging | within 72 hours after extubation
  Number of chest X-rays and NPLUS within 72 hours after extubation
Number of lung imaging based interventions | within 72 hours after extubation
  Number and time points of chest X-ray or NPLUS based interventions
Recruitment maneuvers | within 72 hours after extubation
  Number and time points of recruitment maneuvers (PEEP increase, positioning)
Time to detect consolidations | within 72 hours after extubation
  Time to detect impairment of lung aeration (consolidations)
Lung ultrasound scores (LUS) | up to 24 hours after extubation
  LUS at time point T0 (prior to extubation), T1 (2-4 hours post extubation) and time point T2 (16-24 h post extubation)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Schwaberger, MD PhD, Principal Investigator — Division of Neonatology, Medical University of Graz, Austria
Locations (1):
- Department of Pediatrics, Division of Neonatology, Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided